CLINICAL TRIAL: NCT06957717
Title: Effect of Cow's Milk Kefir on Short Chain Fatty Acid (SCFA), Haemoglobin, and Ferritin Levels of Anemic Adolescent Girls in Yogyakarta, Indonesia
Brief Title: Effect of Cow's Milk Kefir on Short Chain Fatty Acid (SCFA), Haemoglobin, and Ferritin Levels of Anemic Adolescent Girls
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lusyana Gloria Doloksaribu (Other)
Responsible Party: Sponsor-Investigator, Lusyana Gloria Doloksaribu, doctoral students of the faculty of medicine, public health and nursing, Gadjah Mada University, Gadjah Mada University
Organization: Gadjah Mada University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GadjahMada
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiency Anemia
Keywords: Kefir; Short Chain Fatty Acid; Hemoglobin; Ferritin; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Milk; Control Groups

STUDY DESIGN:
Intervention Model Description: Its research is an experimental study, with a Randomized Controlled Trial (RCT) design, pre-posttest design, involving research subjects of adolescent girls (15-18 years) with mild and moderate anemia, at SMKN 1, 2, and 3 Kasihan, Bantul Regency, Yogyakarta, as many as 80 students. Subjects were divided into 2 groups, namely group 1 (treatment group), which was given 120 ml of cow's milk kefir every day and TTD 1 grain/week, and group 2 (control group), which was given 120 ml of cow's milk every day and TTD 1 grain/week. The duration of administration was 2 months. The study outcomes were Short Chain Fatty Acid (SCFA) levels in feces by Gas Chromatography-Mass Spectrometry (GC-MS) method, hemoglobin by Hematology Analyser method, and serum ferritin by Ferritin ELISA measured at the beginning and end of the study. Statistical analysis included univariate, bivariate, and multivariate analysis. Clinical analysis was also conducted to estimate the effect size of the treatment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In addition to participants, service providers, and outcomes assessors, it is also disguised from statisticians or data processors so that the data obtained does not become biased
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Fresh cow's milk drink pasteurized at 72 °C, and fermented by kefir grain (5%) for 24 hours at 25 °C, then filtered to produce cow's milk kefir, and stored at 4 °C for 24 hours before drinking, given as 1 bottle/day of 120 ml + 10% liquid sugar for 2 months.
  Interventions: Combination Product: cow's milk kefir
- control group (Placebo Comparator): Fresh cow's milk drink pasteurized at 72 °C, without fermentation, given 1 bottle/day of 132 ml for 2 months
  Interventions: Combination Product: pasteurized cow's milk

INTERVENTIONS:
Combination Product: cow's milk kefir — group given cow's milk kefir and blood supplement tablets (TTD)
  Other Names: intervention group
  Arms: intervention group
Combination Product: pasteurized cow's milk — group given pasteurized cow's milk and blood supplement tablets (TTD)
  Other Names: control group
  Arms: control group

SUMMARY:
Introduction: The prevalence of anemia among adolescent girls in Indonesia is still quite high. According to the Indonesian Health Survey (IHS) in 2023, it was 18% and is still a national problem. Long-term supplementation of blood supplement tablets (TTD) as an effort made by the government to prevent/overcome anemia has caused side effects, namely dysbiosis by pathogenic bacteria. Giving cow's milk kefir containing various probiotics can overcome the side effects of supplementation, and its metabolites accelerate iron absorption so that iron status in the blood increases and ultimately restores anemia in adolescent girls. Method: It's research is an experimental study, with a Randomized Controlled Trial (RCT) design, pre-posttest design, involving research subjects of adolescent girls (15-18 years) with mild and moderate anemia, at SMKN 1, 2, and 3 Kasihan, Bantul Regency, Yogyakarta as many as 80 students. Subjects were divided into 2 groups, namely group 1 (treatment group), which was given 120 ml of cow's milk kefir every day and TTD 1 grain/week, and group 2 (control group), which was given 120 ml of cow's milk every day and TTD 1 grain/week. The duration of administration was 2 months. The study outcomes were Short Chain Fatty Acid (SCFA) levels in feces by Gas Chromatography-Mass Spectrometry (GC-MS) method, hemoglobin by Hematology Analyser method, and serum ferritin by Ferritin ELISA measured at the beginning and end of the study. Statistical analysis included univariate, bivariate, and multivariate analysis. Clinical analysis was also conducted to estimate the effect size of the treatment

DETAILED DESCRIPTION:
This protocol represents the only doctoral research dissertation proposal I will undertake as part of my dissertation, which does not exist.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls aged 15-18 years
* Have a mild and moderate degree of anemia (Hb 8-11.9 g/dl)
* Have a normal menstrual cycle and duration

Exclusion Criteria:

* Suffering from thalassemia, hemosiderosis, blood cancer, and malaria, based on the doctor's diagnosis in the last 3 months
* Taking supplements other than TTD
* Taking antibiotics in the last 3 months
* Suffering from lactose intolerance through interviews

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Adolescent girls as future mothers
Enrollment: 80 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Short Chain Fatty Acid | 2 months after intervention
  SCFA (acetate, propionate, and butyrate) levels in fresh feces of adolescent girls, using the GC-MS (Gas Chromatography-Mass Spectrometry) Method, were measured before (0 months) and after the intervention (2 months), using a ratio scale.
  The examination procedure included collecting feces in the field according to the procedure at https://drive.google.com/drive/folders/1uXklwFuC-1rnQ1Anim86b7-9pqLSheIz. Fresh feces samples were collected immediately, by storing them in a cool box (to maintain the quality of feces so that it remains stable during storage and transportation, and avoid the maturation process that can affect the results of lab tests, so that the results of the lab analysis carried out can be accurate and valid), and then immediately taken to the laboratory to quantify each of the short chain fatty acids (SCFA) in the sample.
hemoglobin | 2 months after intervention
  Adolescent girls' hemoglobin values in the blood taken from the median cubital vein, using the hematology analyzer method (unit g/dl), were measured before (0 months) and after the intervention (2 months), using a ratio scale.
Ferritin | 2 months after intervention
  Ferritin content in the blood of adolescent girls taken from the median cubital vein, using the Ferritin ELISA method (unit µg/L), was measured before (0 months) and after the intervention (2 months), using a ratio scale

SECONDARY OUTCOMES:
Nutrient intake | 2 months after intervention
  The amount of nutrients iron, folic acid, protein, vitamin C, zinc, energy and fat that enter the body of adolescent girls per day obtained from food and beverages, using the Food Record method carried out for 3 days, consisting of 2 times weekday and 1 time weekend, analyzed using the Nutrisurvey 2007 application, measured before (0 months) and after the intervention (2 months), using a ratio scale.
Nutritional status of adolescent girls (body mass index / age) | 2 months after intervention
  The Z-score or standard deviation (SD) value of adolescent girls after calculating the ratio of body weight in kilograms (kg) squared with height in meters (m) correlated with age, was analyzed using the WHO AnthroPlus application, measured before (0 months) and after the intervention (2 months), using a ratio scale.
  Weight values were obtained by weighing adolescent girls using digital scales with an accuracy of 0.1 kg. Height values were obtained by measuring the height of adolescent girls using a microtoise with an accuracy of 0.1 cm, and age was obtained by asking about the date/month/year of birth of adolescent girls. Using a questionnaire.
Menstrual cycle and duration of adolescent girls | 2 months after intervention
  The physiological process experienced by adolescent girls, namely periodic bleeding from the uterus accompanied by the release of the endometrial wall every month, was obtained through a questionnaire, using an ordinal scale, with the categories (1). Normal if the menstrual cycle ranges from 21-35 days, and the length of menstruation is 3-7 days, and (2). Abnormal if the menstrual cycle ranges <21 days and >35 days, and the duration of menstruation is <3 days and >7 days
Diarrhea | 2 months after intervention
  Complaints of watery or loose bowel movements that occur more than 3 times a day were obtained through a questionnaire, using an ordinal scale, with the categories (1). No diarrhea if the frequency of bowel movements ranged from 1-2 times/day, with a solid consistency, and (2). Diarrhea, the frequency of bowel movements ranging ≥3 times/day, watery, thin consistency

CONTACTS AND LOCATIONS:
Locations (1):
- Gadjah Mada University, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
IPD data will be shared, but in the form of coding.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD can be obtained after the dissertation is registered at the Universitas Gadjah Mada Library or the Faculty of Medicine, Public Health, and Nursing Library
Access Criteria: Only investigator
URL: https://lib.ugm.ac.id/